CLINICAL TRIAL: NCT06721390
Title: Impact of Music Improvisation Training on Cognitive Function in Older Adults
Brief Title: Music Improvisation Training on Cognitive Function in Older Adults
Acronym: Music Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 4R33AG073669-03 (NIH); R33AG073669 (NIH)
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Aging; Cognitive Aging; Cognitive Impairment; Cognitive Training; Mild Cognitive Impairment; Cognitively Normal Older Adults
Keywords: Aging; Brain Aging; Cognition; Cognitive Engagement; Mild Cognitive Impairment; Music; Music-based Intervention; Music Training; Older Adults
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Parallel Assignment - We will conduct a 2-arm randomized controlled trial.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Piano Improvisation (Experimental): This intervention will involve group piano improvisation training sessions once a week for 12 weeks, in addition to daily in-home practice for 4-5 days.
  Interventions: Behavioral: Piano Improvisation
- Music Listening (Active Comparator): The music listening condition will involve group music listening sessions (led by a trained instructor) once a week for 12 weeks and daily in-home music listening practice.
  Interventions: Behavioral: Music Listening

INTERVENTIONS:
Behavioral: Piano Improvisation — Piano Improvisation taught by a professional instructor for 12 weeks.
  Arms: Piano Improvisation
Behavioral: Music Listening — Music Listening facilitated by a professional instructor for 12 weeks.
  Arms: Music Listening

SUMMARY:
This project will study the effects and mechanisms of a music improvisation training intervention on self-regulation of older adults with and without MCI. The investigator's overall hypothesis is that improvisation training will lead to improvements in self-regulation, compared to controls, and that improvisation training will be associated with specific changes in prefrontal brain networks and ultimately cognitive engagement.

DETAILED DESCRIPTION:
Approximately 5.8 million adults age 60 and over in the United States live with Alzheimer disease and related dementias (AD/ADRD) at a cost of $290 billion per year. Older adults with mild cognitive impairment (MCI), an intermediate stage between typical aging and dementia, are 3-5 times more likely to progress to AD than those with normal cognition. Late-life engagement in cognitively challenging activities is associated with decreased risk of cognitive decline, and there is a need to address cognitive inactivity. Music interventions are a promising strategy to address late-life cognitive inactivity. Music training can change brain structure and function in non-musician adults, thereby leading to cognitive, perceptual, and psychosocial advantages. These changes in cognitive function are thought to occur because the multimodal, complex nature of music facilitates training-induced neural plasticity. However, the mechanisms are not yet understood, and most studies used traditional or rote keyboard training techniques. Music training based on improvisation principles-the spontaneous generation of musical melodies and rhythms-will likely have more potent effects on cognition and brain function. Improvisation facilitates cognitive flexibility, self-monitoring, novel idea generation, execution of unplanned motor sequences and entrance into a state of flow. Biologically, improvisation is associated with distinct neural patterns involving activation of prefrontal networks and other brain networks that are affected by aging. As a mechanism of behavior change, it is likely that improvisation training will uniquely improve self-regulation (the ability to monitor and control one's own behavior, emotions, or thoughts and modify to situational demands). Yet, no research has tested whether improvisation training can improve self-regulation and facilitate maintenance of cognitively challenging activities among older adults with and without MCI. This project will develop and test the effects and mechanisms of a music improvisation training intervention on self-regulation of older adults with and without MCI. Our overall hypothesis is that improvisation training will lead to improvements in self-regulation, compared to controls, and that improvisation training will be associated with specific changes in prefrontal brain networks and ultimately cognitive engagement. Our project has two phases. In the R61 phase, the study will develop a music improvisation training intervention that aims to improve self-regulation among older adults with and without MCI and conduct a 2-arm randomized pilot study to (i) examine feasibility and acceptability of the intervention and study methods and (ii) determine its effects on the hypothesized mechanism of self-regulation. If milestones are met, the study will proceed to the R33 phase and conduct a randomized mechanistic trial to examine the effects of the intervention, compared to an attention control, on self-regulation and cognitive engagement among older adults with and without MCI. The findings from this study will improve our understanding of the underlying mechanisms of how music training interventions can facilitate behavior change to maintain health of older adults.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 and over
* Living independently in the community
* Sufficient visual and hearing acuity (age-related to normal hearing loss, with assistive devices) as measured by audiometer
* Less than three years of formal music training (as indicated by private music lessons does not include group or ensemble classes) and not currently reading or engaging in music performance
* English fluency rated fairly well to well
* MoCA score of 22-30 or diagnosis of "mild cognitive impairment
* Not currently taking psychoactive medications, antidepressants, or sleep medications that could adversely affect cognitive abilities.

Exclusion Criteria:

* Medical diagnosis of dementia (any etiology)
* Inability to move the hands or use all 10 digits (extensive arthritis, neuropathy, missing digits)
* Score < 22 on MoCA
* Current (but not prior) severe psychiatric disorder, serious medical condition (e.g., stroke, TIA) that would interfere with participation in the study
* Poor English fluency
* Musician or previously trained in jazz improvisation, more than three years of formal music instruction or training and/or currently engaged in musical performance
* Plans to move out of the area within six months

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Florida Cognitive Activities Scale | Baseline and 12-week Post Intervention
  The Florida Cognitive Activities Scale is a 25-item scale (0-never to 5-daily) used to assess the cognitive activity in elderly populations. There are two subscales, the Higher Cognitive Abilities and Frequent Cognitive Abilities, and also a measure of self-reported maintenance of cognitive activity
Short Self Regulatory Questionnaire | Baseline and 12-week Post Intervention
  Self-report measure of the ability to regulate one's behavior in a goal-oriented way. This self-reported questionnaire contains 31 items, each item was scored on a five-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). The questionnaire scores ranged from 31 to 155, with higher scores indicating better self-regulation behavior

SECONDARY OUTCOMES:
National Institutes of Health ToolBox Self-Efficacy | Baseline and 12-week Post Intervention
  The NIH Toolbox Self-Efficacy Scale is a 10-item self-reported measure that assesses belief in one's capacity to manage and have control over meaningful events in life. Scores for each item range from 1 to 5 (never to very often).
  Higher scores indicate higher self-efficacy.
Short GRIT Scale | Baseline and 12-week Post Intervention
  The Grist-S is a self-report, 8-item questionnaire that measures the extent to which individuals are able to maintain focus and interest and persevere in obtaining long-term goals. Scores for each item range from 1 to 5, with overall scores being calculated by added up all points and dividing by 8. Higher scores indicate a higher level of "grit," or perseverance.
Five Facets of Mindfulness | Baseline and 12-week Post Intervention
  Measures components of mindfulness, which is a tendency to attend to the present moment with a non-judgemental attitude. Scores for each item range from 1 to 6 (never to always true). Mindfulness and self-regulation ability have been identified as closely aligned in recent theoretical frameworks (e.g., the self- awareness, -regulation, and - transcendence model of mindfulness
National Institutes of Health Toolbox Loneliness Scale | Baseline and 12-week Post Intervention
  Self-report measure that assesses perceptions of loneliness and assesses the extent to which an individual feels alone or socially isolated from other individuals. The NIH Toolbox Loneliness Survey is a self-report measure that assesses perceptions of loneliness using a 5-item fixed length form.
National Institutes of Health Toolbox Apathy | Baseline and 12-week Post Intervention
  National Institutes of Health Toolbox Apathy Instruments measuring deficits in-goal directed behavior and decrements in in-goal related thought content. It is 7 items, each item is scored on a 4-point Likert scale (not at all true to very true). The total score ranges from 18 to 72, with higher scores indicating more apathy.
Geriatric Depression Scale - Short Form | Baseline and 12-week Post Intervention
  A short form comprising of 15-items, which is effective for the diagnosis of depression of elderly, is more simple, brief and time-effective.
10-item Personality Inventory | Baseline and 12-week Post Intervention
  Brief assessment of the Big Five Personality Dimensions: 1. Extraversion, 2. Agreeableness, 3. Conscientiousness, 4.
  Emotional Stability, and 5. Openness to Experience consisting of 10 items. Scores range from 1 (disagree strongly) to 7 (agree strongly).

CONTACTS AND LOCATIONS:
Overall Officials: Julene Johnson, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- The study is taking place at community sites in San Francisco., San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No